CLINICAL TRIAL: NCT05204589
Title: Heterologous Prime-boost Immunization with an Aerosolised Adenovirus Type-5 Vector-based COVID-19 Vaccine (Ad5-nCoV) After Two-dose Priming with an Inactivated SARS-CoV-2 Vaccine in Adults Aged 18 Years and Above: a Multicenter, Open-label, Partially Parallel-controlled Clinical Trial
Brief Title: Heterologous Boost Immunization with an Aerosolised Ad5-nCoV After Two-dose Priming with an Inactivated SARS-CoV-2 Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Anhui Provincial Center for Disease Control and Prevention (Unknown); Shandong Province Centers for Disease Control and Prevention (Other); Hunan Provincial Center for Disease Control and Prevention (Other); Yunnan Center for Disease Control and Prevention (Other); Chongqing Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT137
Record Dates: First submitted 2022-01-21; First posted 2022-01-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Aerosolised COVID-19 vaccine; Recombinant Ad5 Vector; Inactivated Vaccine; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Subjects in safety cohort will receive one heterologous booster dose of aerosolized Ad5-nCoV
  Interventions: Biological: Aerosolized Ad5-nCoV
- Group B (Experimental): Subjects in immunogenicity cohort will receive one heterologous booster dose of aerosolized Ad5-nCoV
  Interventions: Biological: Aerosolized Ad5-nCoV
- Group C (Experimental): Subjects in immunogenicity cohort will receive one homologous booster dose of ICV.
  Interventions: Biological: Inactivated SARS-CoV-2 vaccine

INTERVENTIONS:
Biological: Aerosolized Ad5-nCoV — Aerosolized Ad5-nCoV is produced by CanSino Biologics Inc. It is a liquid dosage form, 0.1 ml / dose, contains 1×10^10 virus particles of recombinant replication defective human type 5 adenovirus expressing SARS-CoV-2 S protein, aerosol inhalation.
  Arms: Group A; Group B
Biological: Inactivated SARS-CoV-2 vaccine — Inactivated SARS-CoV-2 vaccine is homologous to the priming series which have been administered to the subjects, produced by SinoVac Biotech Co,. Ltd, Beijing Institute of Biological Products Co,. Ltd, Wuhan Institute of Biological Products Co,. Ltd, or Biokangtai.
  Arms: Group C

SUMMARY:
This is a multicenter, open-label, partially radomized, parallel-controlled clinical trial to evaluate the safety and immunogenicity of heterologous prime-boost immunization with an aerosolised adenovirus type-5 vector-based COVID-19 vaccine (Ad5-nCoV-IH) after two-dose priming with an inactivated SARS-CoV-2 vaccine (ICV) in adults aged 18 years and above. 10420 healthy subjects aged over or equal to 18 years whom have received two doses of ICV before 6 months or more, will be recruited from six provinces in China in this study.Of them, 10000 eligible participants in an open cohort will receive a booster dose of Ad5-nCoV-IH to evaluate the safety profile. Another 420 participants were involved in immunogenicity cohort and randomized in a ratio of 1:1 to receive a boost of Ad5-nCoV-IH or ICV. The ICV homologous to the priming series will be supplied as the booster. The occurrence of adverse reactions within 28 days and serious adverse events within 6 months after vaccination will be observed in all participants. In addition, blood and saliva samples will be collected from all participants in immunogenicity cohort on the day 0 before and 14, 28 and month 3 and 6 after the booster vaccination. Each subject will remain in this study for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Health subjects aged ≥18 years.
* Have received two-dose inactivated SARS-CoV-2 vaccine before 6 months or more.
* The subject can provide with informed consent and sign informed consent form (ICF).
* The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the 6-month follow-up of the study.

Exclusion Criteria:

* Have the medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* Be allergic to any component of the research vaccines, or used to have a history of hypersensitivity or serious reactions to vaccination.
* Women with positive urine pregnancy test.
* Have acute febrile diseases and infectious diseases.
* Axillary temperature>37.0℃.
* Have serious cardiovascular disease, such as arrhythmia, conduction block, myocardial infarction, severe hypertension that cannot be controlled by medication (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg when measured in the field).
* Have severe chronic diseases or condition in progress cannot be smoothly controlled, such as asthma, diabetes, thyroid disease.
* Congenital or acquired angioedema / neuroedema.
* Have the history of urticaria 1 year before receiving the investigational vaccine.
* Have asplenia or functional asplenia.
* Patients with chronic obstructive pulmonary disease, pulmonary fibrosis and other pulmonary abnormalities.
* Have history of SARS-CoV-2 infection or COVID-19.
* Have symptoms of upper respiratory tract infection.
* Have traveled to medium or high risk areas or traveled abroad in the past 21 days, and epidemiologically contacted with SARS-CoV-2.
* Any medical, psychological, social, or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10285 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions within 28 days after the booster dose. | Within 28 days the booster dose
  Incidence of adverse reactions within 28 days after the booster dose.
GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose in immunogenicity cohort. | On day 28 after the booster dose
  GMT of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose in immunogenicity cohort.

SECONDARY OUTCOMES:
Incidence of adverse reactions within 30 minutes after the booster dose. | Within 30 minutes after the booster dose
  Incidence of adverse reactions within 30 minutes after the booster dose.
Incidence of adverse reactions within 14 days after the booster dose. | Within 14 days after the booster dose
  Incidence of adverse reactions within 14 days after the booster dose.
Incidence of adverse events within 28 days after the booster dose. | Within 28 days after the booster dose
  Incidence of adverse events within 28 days after the booster dose.
Incidence of serious adverse events (SAE) till the 6 months after the booster dose. | Within 6 months after the booster dose
  Incidence of serious adverse events (SAE) till the 6 months after booster vaccination.
Fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose. | On day 28 after the boost vaccination
  Fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 28 after the booster dose in immunogenicity cohort.
GMT, Fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus on day 14, month 3 and 6 after the booster dose. | On day 14, month 3 and 6 after the booster dose
  GMT, Fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus as compared to baseline on day 14, month 3 and 6 after the booster dose.
GMT, fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus at month 3, 6, and 12 after the booster dose. | At month 3, 6, and 12 after the boost vaccination.
  GMT, fold increase and seroconversion of neutralizing antibodies against live SARS-CoV-2 virus at month 3, 6, and 12 after the booster dose.
Geometric mean concentration (GMC), fold increase and seroconversion of binding IgG against S protein of SARS-CoV-2 on day 14, day 28 and month 3 and 6 after the booster dose. | On day 14, day 28 and month 3 and 6 after the booster dose
  Geometric mean concentration (GMC), fold increase and seroconversion of binding IgG against S protein of SARS-CoV-2 on day 14, day 28 and month 3 and 6 after the booster dose.
GMT of neutralizing antibodies against live SARS-CoV-2 virus in participants with pre-existing anti-Ad5 antibody titers>1:200 or ≤1:200 at baseline. | On day 28 after the booster dose
  GMT of neutralizing antibodies against live SARS-CoV-2 virus in participants with pre-existing anti-Ad5 antibody titers>1:200 or ≤1:200 at baseline.
GMT, fold increase and seroconversion of neutralizing antibodies against VOC/VOI of SARS-CoV-2 virus on day 28 after the booster dose. | On day 28 after the booster dose
  GMT, fold increase and seroconversion of neutralizing antibodies against VOC/VOI of SARS-CoV-2 virus on day 28 after the booster dose.
The levels of IFN-γ、TNF-α、IL-2、IL-4、IL-5、IL-13 secreted by specific T cells on day 14 after the booster vaccination. | On day 14 after the booster vaccination
  The levels of IFN-γ、TNF-α、IL-2、IL-4、IL-5、IL-13 secreted by specific T cells on day 14 after the booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Prof, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Li JX, Hou LH, Gou JB, Yin ZD, Wu SP, Wang FZ, Zhang Z, Peng ZH, Zhu T, Shen HB, Chen W, Zhu FC; Six-Province COVID-19 Vaccine Study Group. Safety, immunogenicity and protection of heterologous boost with an aerosolised Ad5-nCoV after two-dose inactivated COVID-19 vaccines in adults: a multicentre, open-label phase 3 trial. Lancet Infect Dis. 2023 Oct;23(10):1143-1152. doi: 10.1016/S1473-3099(23)00350-X. Epub 2023 Jun 20. PMID 37352880